CLINICAL TRIAL: NCT06006429
Title: Digital Extraction and Scientific Visualization of Clinical Characteristics From 3D Data From Intraoral Scanners for Dental and Periodontal Pathologies Research : Computer Formalization and Feasibility Study
Brief Title: Intraoral Scanners as Periodontal and Dental Pathologies Diagnosis Tools
Acronym: Odonto3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PO21146
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis; Gingivitis; Dental Caries; Diagnosis
Keywords: Periodontal diseases; Dental caries; intra-oral camera; diagnosis
MeSH Terms: conditions — Periodontitis; Gingivitis; Dental Caries; Disease; Periodontal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Numerical dental impression by intraoral scanner

INTERVENTIONS:
Other: Numerical dental impression by intraoral scanner — Intervention consists in an 3D intra oral representation of the oral cavity

SUMMARY:
Periodontal diseases and dental pathologies are highly prevalent oral diseases. Thirty-three to fifty percent of adult population presented at least one untreated caries and more than 50% of French population are affected by severe periodontitis. These diseases affect dental organ or periodontal attached system but could have negative impact on general health, quality of life, word and individual well-being. Association between chronic diseases as diabetes, rheumatoid arthritis, cardiovascular diseases, and oral health have been well investigated. Dental and periodontal diagnosis is dependent of various clinical parameters time consuming and dependent operator. It represents a public health challenge. Informatic analysis detecting diseases could be a time gain and a more precise diagnosis tool. Today, any software or algorithm allow automatized detection, clinical qualitative or quantitative indices recording while these informations are present in numeric models

DETAILED DESCRIPTION:
The present study explores the effectiveness of intraoral scanners in the field of dental caries and periodontal diseases diagnosis Patients presenting at least on recession are recruited without randomization. A clinical examination is performed, and a 3D impression of their mouth is obtained by intraoral scanners.

The investigators hypothesized that the 3D intra oral representations could improve oral diagnosis in patients compared to clinical examination in term of time consummation and precision. In a first time, this could be achieved by the comparison of the recession measurement obtained by a clinical measure (Ramfjord, 1959) or obtained by artificial intelligence.

The secondary objectives are :

* To compare clinical and numerical dento-prosthetic diagram
* To compare clinical and numerical plaque control record index (O'Leary et al., 1973)
* To compare clinical and numerical Decayed, Missed and Filled Teeth index (Klein and Palmer, 1940)
* To compare clinical and numerical detection of mucosal lesions

ELIGIBILITY:
Inclusion Criteria:

* adultes
* consulting the Dental Care Service of the university hospital of Reims
* presenting at least one gingival recession
* presenting at least 10 pairs of opposing teeth
* speaking French
* who signed the informed consent form
* affiliated to the French Social Security system

Exclusion Criteria:

Patients presenting :

* pregnancy or breastfeeding
* orthodontic treatments
* patients under legal protection, trusteeship or guardianship
* unable to understand auto-questionnary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Recession measurement concordance (Ramfjord, 1959) | Day 1
  Recession depths is measured between the cementum-enamel junction and the edge of the marginal gingiva.
  The clinical and numerical scored will be compared.

SECONDARY OUTCOMES:
Dento-prosthetic diagram concordance | Day 1
  Recording the presence or absence of tooth The clinical and numerical scored will be compared.
Plaque Control Record Concordance (O'Leary et al., 1972) | Day 1
  Plaque control record will be recorded on individual tooth surfaces (mesial, distal, facial, lingual).
  PCR is calculated according the following formula :
  PCR = (Number of faces with plaque / Total number of faces) x 100
  The clinical and numerical scored will be compared.
Gingival Index Concordance (Loe and Silness, 1963) | Day 1
  Gingival index is scored as described :
  0 Normal gingival Natural coral pink gingival with no inflammation
  1. Mild inflammation Slight changes in color, slight edema. No bleeding on probing
  2. Moderate inflammation Redness, edema and glazing Bleeding under probing
  3. Severe inflammation Marked redness and edema/ulceration Tendency to bleed spontaneously
  The clinical and numerical scored will be compared.
Decayed, Missed and Filled Teeth Index (Klein and Palmer, 1940) | Day 1
  DMFT is the sum of decayed, missed due to caries and filled teech in the permanent teeth.
  Third molars are excepted.
  The clinical and numerical scored will be compared.
Mucosal lesions detection | Day 1
  Presence or absence of mucosal lesions.
  The clinical and numerical lesions will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France